CLINICAL TRIAL: NCT01450293
Title: Safety and Immunogenicity of Heterologous Prime-boost Vaccination With the Candidate Malaria Vaccines AdCh63 ME-TRAP and MVA ME-TRAP in Healthy Infants in a Malaria- Endemic Area
Brief Title: AdCh63 ME-TRAP and MVA ME-TRAP Malaria Vaccines Evaluation in Healthy Children in a Malaria Endemic Area
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VAC042
Record Dates: First submitted 2011-10-03; First posted 2011-10-12 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Malaria
Keywords: Immune response
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group A (Experimental): 5 to 12 months old infants; AdCh63 ME-TRAP, MVA ME-TRAP
  Interventions: Biological: AdCh63 ME-TRAP, MVA ME-TRAP
- Group B (Experimental): 5 to 12 months old infants; AdCh63 ME-TRAP, MVA ME-TRAP
  Interventions: Biological: AdCH63 ME-TRAP, MVA ME-TRAP
- Group C (No Intervention): 5 to 12 months old infants; no vaccination
- Group D (Experimental): 10 week old babies; AdCh63 ME-TRAP, MVA ME-TRAP
  Interventions: Biological: AdCh63 ME-TRAP, MVA ME-TRAP
- Group E (Experimental): 10 week old babies; AdCh63 ME-TRAP, MVA ME-TRAP
  Interventions: Biological: AdCH63 ME-TRAP, MVA ME-TRAP
- Group F (No Intervention): 10 week old babies; no vaccination

INTERVENTIONS:
Biological: AdCh63 ME-TRAP, MVA ME-TRAP — 1x10^10 vp AdCH63 ME-TRAP followed by 1x10^8 pfu MVA ME-TRAP 8 weeks later. Intramuscular needle injection into the anterolateral thigh.
  Arms: Group A; Group D
Biological: AdCH63 ME-TRAP, MVA ME-TRAP — 5x10^10 vp AdCH63 ME-TRAP followed by 1x10^8 pfu MVA ME-TRAP 8 weeks later. Intramuscular needle injection into the anterolateral thigh.
  Arms: Group B; Group E

SUMMARY:
Infants in malaria-endemic regions of Africa are an important target for vaccination against malaria in view of the enormous disease burden of malaria in this population. The purpose of this trial is to assess the safety and immunogenicity of MVA ME-TRAP and AdCH63 ME-TRAP candidate vaccines in healthy children in a malaria endemic region. The regimen proposed here has protected non-immune volunteers in Oxford against sporozoite challenge, and so may be protective against naturally acquired infection in the Gambia. Administration of AdCh63 ME-TRAP and MVA ME-TRAP to infants in this study will occur at intervals of at least two weeks from the administration of routine infant immunisations, given according to the Gambian EPI.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants aged 10 weeks and 5-12 months at the time of enrollment with consenting parents.

Exclusion Criteria:

* Clinically significant history of skin disorder (psoriasis, contact dermatitis etc.), allergy, symptomatic immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurological illness.
* Severe malnutrition.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines, e.g. egg products, Kathon, neomycin, betapropiolactone.
* History of splenectomy Haemoglobin less than 8.0 g/dL, where judged to be clinically significant in the opinion of the investigator
* Serum Creatinine concentration greater than 70 mol/L, where judged to be clinically significant in the opinion of the investigator
* Serum ALT concentration greater than 45 U/L, where judged to be clinically significant in the opinion of the investigator
* Blood transfusion within one month of enrollment.
* History of vaccination with previous experimental malaria vaccines. -Administration of any other vaccine or immunoglobulin less than two weeks before vaccination with the IMPs Current participation in another clinical trial, or within 12 weeks of this study.
* Any other finding which in the opinion of the investigators would increase the risk of an adverse outcome from participation in the trial.
* Likelihood of travel away from the study area
* Maternal HIV infection Positive malaria antigen test at screening
* Failure to have received, prior to enrollment, the routine EPI vaccinations due according to the Gambian EPI schedule.

Ages: 10 Weeks to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2011-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety of heterologous prime-boost vaccination with AdCh63 ME-TRAP followed eight weeks later by MVA ME-TRAP | Participants will be followed for the duration of the study, an expected average of 16 months
  To assess the safety of heterologous prime-boost vaccination of healthy infants in a malaria-endemic area with AdCh63 ME-TRAP followed eight weeks later by MVA ME-TRAP by recording local and systemic solicited and unsolicited adverse events

SECONDARY OUTCOMES:
Immunogenicity of heterologous prime-boost vaccination with AdCh63 ME-TRAP followed eight weeks later by MVA ME-TRAP | Participants will be followed for the duration of the study, an expected average of 16 months
  To assess the immunogenicity of heterologous prime-boost vaccination of healthy infants in a malaria-endemic area with AdCh63 ME-TRAP followed eight weeks later by MVA ME-TRAP by assessing induced antibody and T cell response to the vaccine insert

CONTACTS AND LOCATIONS:
Overall Officials: Kalifa Bojang, Principal Investigator — Medical Research Council PO Box 273, Banjul The Gambia
Locations (1):
- Medical Research Council Laboratories, Banjul, The Gambia